CLINICAL TRIAL: NCT04481594
Title: A Randomized, Double-Blind, Placebo Controlled, Sequential Parallel Group, Single and Multiple Ascending Doses (SAD/MAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HPN-01
Brief Title: A Study to Evaluate the Safety and Tolerability of Single and Multiple Ascending Doses of HPN-01 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hepanova Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HPN-01-US-101
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: double-blind (participant, investigator)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HPN-01 (Experimental): Part 1: Including 6 dose cohorts (25 mg, 50 mg, 100 mg, 150 mg, 200 mg and 300 mg). Each dose cohort will receive a single dose of HPN-01. One cohort of Part 1 will receive HPN-01 after a standard high fat/high calorie breakfast (the fed condition) to investigate the effect of food on the pharmacokinetics of HPN-01.
  Part 2: Including 3 dose cohorts (50 mg, 100 mg and 200 mg). Each dose cohort will receive HPN-01 once daily for a consecutive 14 days.
  Interventions: Drug: HPN-01
- Placebo (Placebo Comparator): Part 1: Including 6 dose cohorts (25 mg, 50 mg, 100 mg, 150 mg, 200 mg and 300 mg). Each dose cohort will receive a single dose of HPN-01 placebo.
  Part 2: Including 3 dose cohorts (50 mg, 100 mg and 200 mg). Each dose cohort will receive HPN-01 placebo once daily for a consecutive 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPN-01 — 25 mg, 50 mg, 100 mg, 150 mg, 200 mg and 300 mg HPN-01 capsules
  Arms: HPN-01
Drug: Placebo — 25 mg, 50 mg, 100 mg, 150 mg, 200 mg and 300 mg HPN-01 placebo capsules
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled first-in-human study in which the safety, tolerability, pharmacokinetics and pharmacodynamics of orally administered HPN-01 will be evaluated in healthy subjects

DETAILED DESCRIPTION:
This study aims to obtain safety, tolerability, pharmacokinetic and pharmacodynamic data when HPN-01 is orally administered as single doses and as multiple doses to healthy subjects.

The study will be conducted in 2 parts: a single ascending dose (SAD) phase (Part 1) and a multiple ascending dose (MAD) phase (Part 2). One cohort of Part 1 will receive HPN-01 after a standard high fat/high calorie breakfast (the fed condition) to investigate the effect of food on the pharmacokinetics of HPN-01.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 55 years, inclusive;
3. Female subjects have a negative pregnancy test result at screening and admission to the study site, and meet one of the following criteria:

   1. Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Surgically sterile for at least 3 months prior to screening by one of the following means:

      * Bilateral tubal ligation
      * Bilateral salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   3. Postmenopausal, defined as the following:

      * Last menstrual period greater than 12 months prior to screening
      * Postmenopausal status confirmed by serum FSH and estradiol levels at screening;
4. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
5. Normal renal function (eGFR > 90 ml/min/1.75 m2) as determined by Investigator following review of clinical laboratory test results;
6. Non-smoker and has not been exposed to any products containing nicotine in the last 6 months;
7. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center;
9. Male subjects must agree to utilize a highly effective method of contraception (condom plus spermicide) during heterosexual intercourse from clinic admission until 12 weeks following the end of study visit;
10. Male subjects with female partners of child-bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Known or suspected malignancy;
3. Reported history of pancreatitis or gall stones;
4. Reported history of unexplained syncope, symptomatic hypotension or hypoglycemia;
5. Family history of long QTc syndrome;
6. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
7. Poor venous access;
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B core (IgG and IgM) and surface antigen (HBsAg), Hepatitis A antibody (IgM), hepatitis C antibody (IgG), or hepatitis E (IgG and IgM) at Screening;
9. Donated or lost >500 mL of blood in the previous 3 months prior to screening;
10. Taken an investigational drug or participated in a clinical trial within 3 months (or 5 half-lives) prior to first dose of study drug, whichever is longer;
11. Taken any prescription medications (with the exception of hormonal contraceptive) within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
12. Hospital admission or major surgery within 6 months prior to screening;
13. A history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
14. A history of alcohol abuse according to medical history (≥ 2 drinks per day for male and ≥ 1 drink per day for female) within 9 months prior to screening;
15. A positive screen for alcohol, drugs of abuse at screening or admission;
16. An unwillingness or inability to comply with food and beverage restrictions during study participation;
17. Use of over-the-counter (OTC) medication within 7 days, and/or herbal medications (including St John's Wort, herbal teas, garlic extracts) within 7 days prior to first dose of study drug (Note: Use of acetaminophen at < 2 g/day is permitted until 24 hours prior to dosing);
18. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Single-dose PK Parameter | Up to 72 hours postdose
  Cmax of HPN-01
Single-dose PK Parameter | Up to 72 hours postdose
  AUClast of HPN-01
Single-dose PK Parameter | Up to 72 hours postdose
  AUCinf of HPN-01
Multiple-dose PK Parameters | Up to 24 hours postdose
  Cmax of HPN-01
Multiple-dose PK Parameters | Up to 24 hours postdose
  Ctau of HPN-01
Multiple-dose PK Parameters | Up to 24 hours postdose
  AUCtau of HPN-01
Incidence of Adverse Events | Up to 15 days plus 6 days
Proportion of Participants with 12-lead ECG Abnormalities | Up to 15 days plus 6 days
Proportion of Participants with Clinical Laboratory Abnormalities | Up to 15 days plus 6 days

SECONDARY OUTCOMES:
Measurement of PD Biomarker Level of Fibroblast Growth Factor 19 (FGF19) Following Oral Single and Multiple Ascending Dose Administration | Up to 24 hours postdose
Measurement of PD Biomarker Level of C4 Following Oral Single and Multiple Ascending Dose Administration | Up to 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services, Inc, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No